Study Title: Whey Protein Support to Metabolic and Performance Adaptations in Response to High Intensity Interval Training in Young Adult Men

NCT: 7867835

Date Last Reviewed by Education & Health Sciences Ethical Committee at University of Limerick: 20<sup>th</sup> December 2017

Uploaded: 29th June 2018



# **Participant Information Sheet**

Title of Study: Whey Protein Support to Metabolic and Performance Adaptations in Response to High Intensity Interval Training in Young Adult Men

You are being invited to participate in a study at the University of Limerick investigating the effects of HIIT on your metabolism, cognitive function, mood and performance. This information sheet will inform you about the study.

#### What is the study about?

This study aims to examine how attention toward positive or negative images may be associated with your mood before and after 30-40 minutes of HIIT, and the effects of HIIT on markers of exercise metabolism and performance.

# What will you have to do?

You will be asked to report to the PESS building on 13 occasions totalling an 18-hour commitment.

**Visit 1:** You will be provided with information about all study procedures, risks, and benefits of participation (as outlined in this participant information sheet). Once you feel all your questions about the study have been answered, you will sign an informed consent form to indicate that you understand the study procedures and agree to participate.

You will then complete a series of questionnaires about your physical activity and medical history, your mood, and your cognitive function that will require approximately 20 minutes to complete. You will have your body composition analysed using an electronic scanner and you will then undertake a cycling performance trial lasting approximately 15 minutes. Total time commitment for this visit will be a maximum of 60 minutes.

**Visit 2:** During the second visit, which will be scheduled approximately 48 hours (2 days) following the first visit, you will complete a single Wingate test and two cycling trials, one at below your maximum effort (20 minutes) and one at maximum effort (20 minutes) with 15 minutes rest between each trial. Total time commitment for this visit will be a maximum of 90 minutes.

**Visit 3:** You will attend the lab after an overnight fast and a resting muscle biopsy will be obtained under local anaesthetic. Following this you will consume a supplement or placebo drink ~45 minutes prior to completing 4 bouts of high intensity exercise lasting 30s each with 4 minutes recovery between intervals. Venous blood samples will be collected before and after the exercise session. You will also complete a series of questionnaires about your mood and your cognitive function that will require approximately 20 minutes. A second muscle biopsy will again be obtained under local anaesthetic ~3 hours post-exercise. Total time commitment for this visit will be a maximum of 3 hours.

**Visits 4-10:** You will attend the lab after an overnight fast and consume a supplement or placebo drink ~45 minutes prior to completing 4-6 bouts of high intensity exercise lasting 30s each with 4 minutes recovery between intervals. Total time commitment for this visit will be a maximum of 80 minutes.

Visit 11: You will attend the lab after an overnight fast and consume a supplement or placebo drink ~45 minutes prior to completing 6 bouts of high intensity exercise lasting 30s each with 4 minutes recovery between intervals. You will also complete a series of questionnaires about your mood and your cognitive function that will require approximately 20 minutes. Total time commitment for this visit will be a maximum of 90 minutes.

#### **Visit 12:**

You will attend the lab after an overnight fast and a resting muscle biopsy will be obtained under local anaesthetic, as well as a venous blood sample. You will have your body composition analysed using an electronic scanner. Total time commitment for this visit will be a maximum of 50 minutes.

**Visit 13:** You will complete a Wingate test and two cycling trials similar to visit 2. Total time commitment for this visit will be a maximum of 90 minutes.

#### What are the risks?

There are minimal risks associated with aerobic exercise. Some, but not all, individuals experience shortness of breath, discomfort, and/or soreness during and following HIIT.

### What if I do not want to take part?

Your time and effort is greatly appreciated. If you do not wish to take part it is entirely up to you and this is not a problem. You can withdraw from the study or a part of it at any time without reason or consequence.

### What happens to the information about me that is gathered?

Information obtained about you for this study will be kept confidential and will be stored anonymously on a password protected computer or locked cabinet in the office of the principal investigators. Every effort will be made to maintain the confidentiality of your participation in this project. Each participant's name will be paired with a code number by the principal investigators. This code number will appear on all written and electronic study materials. The list pairing the participant's name to the assigned code number will be kept separate from all research materials and will be available only to the principal investigators. Study data may be used to generate a publication in a scientific journal but all data will be reported as a group and no individual data will be identifiable.

### Who else is taking part?

It is hoped that 39 other volunteers from the University of Limerick staff and student population will complete the study.

### What happens if something goes wrong?

In the unlikely event something goes wrong, testing will cease immediately until normal circumstances are resumed. In the event of an emergency, established University safety procedures will be initiated

What if I have more questions or do not understand something? Please feel free to ask any questions or for further information see contact details below.

### **Contact details**

Dr. Brian Carson

Email: Brian.Carson@ul.ie Phone No.: (061) 234943

OR

Dr. Matthew Herring

Email: Matthew.Herring@ul.ie Phone No.: (061) 234762

Yours sincerely,

Dr Brian Carson, Dr Matthew Herring PESS Department University of Limerick 061-234943; 061-234762

This research study has received Ethics approval from the Education and Health Sciences Research Ethics Committee (). If you have any concerns about this study and wish to contact someone independent you may contact:

Chairman Education and Health Sciences Research Ethics Committee EHS Faculty Office University of Limerick Tel (061) 234101

Email: ehsresearchethics@ul.ie



#### **Participant Informed Consent**

Title of Study: Whey Protein Support to Metabolic and Performance Adaptations in Response to High Intensity Interval Training in Young Adult Men

Should you agree to participate in this study please read the following statements and sign the consent section below.

- I have read and understand the volunteer information sheet.
- I understand what the study is about, and what the results will be used for.
- I understand that what the researchers find out in this study may be shared with others but no identifying information will be given to anyone in any written material.
- I am fully aware of all of the measures involving myself, and of any risks and benefits associated with the study.
- I know that my participation is voluntary and that I can withdraw from the study at any stage without giving any reason.

# For the volunteer

I consent/give permission to my involvement in this research study after agreeing to all of the above statements.

| Name (please print): | |
|---------------------------------------|-------|
| Signature: | Date: |
| Investigator Signature: | Date: |
| Yours sincerely, | |
| Du Drieg Courses Du Matthewelle mises | |

Dr Brian Carson, Dr Matthew Herring PESS Department University of Limerick 061-234943; 061-234762

This research study has received Ethics approval from the Education and Health Sciences Research Ethics Committee (quote approval number). If you have any concerns about this study and wish to contact someone independent you may contact:

Chairman Education and Health Sciences Research Ethics Committee EHS Faculty Office University of Limerick Tel (061) 234101

Email: ehsresearchethics@ul.ie